CLINICAL TRIAL: NCT02641249
Title: Neuromodulation of Limb Proprioceptive Afferents Using a Vibratory Device to Decrease Apnea, Intermittent Hypoxia and Bradycardia of Prematurity.
Brief Title: Non-invasive Intervention for Apnea of Prematurity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Kalpashri Kesavan, Clinical Instructor, University of California, Los Angeles
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB#14-000804
Record Dates: First submitted 2015-12-18; First posted 2015-12-29 (Estimated); Results first posted 2017-05-09 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2016-11

CONDITIONS: Apnea of Prematurity; Hypoxia; Bradycardia
MeSH Terms: conditions — Apnea; Hypoxia; Bradycardia

STUDY DESIGN:
Intervention Model Description: In the same subject there were 2 periods:
  Arm 1. 'No intervention' period (no vibrations) - two 6 hour epochs - total of 12 hours of 'No intervention' Arm 2. Experimental period (with vibrations) - two 6 hour epochs - total of 12 hours of 'vibration intervention'
  In the same subjects cardiorespiratory parameters - heart rate, respiratory rate and oxygen saturation were compared during the experimental period (vibration) and druing the no intervention period (no vibration).
Masking Description: Open Label
Oversight: Data Monitoring Committee: No

ARMS (2):
- No vibration (No Intervention): In the same subject cardiorespiratory parameters - heart rate, respiratory rate and oxygen saturation were compared during the procedure (vibration) and without procedure (no vibration). The same subject had both control and treatment periods.
- Vibration (Experimental): In the same subject cardiorespiratory parameters - heart rate, respiratory rate and oxygen saturation were compared during the procedure (vibration) and without procedure (no vibration). The same subject had both control and treatment periods.
  Interventions: Device: Vibration

INTERVENTIONS:
Device: Vibration — A device providing vibrations is placed on the subject and vibration is turned on and off in a 6 hour on/off sequence. Heart rate, respiratory pauses and oxygen saturation are compared during vibration (intervention) and without vibration (no intervention) in the same subject.
  Other Names: (no generic name)
  Arms: Vibration

SUMMARY:
Purpose of Study: Apnea of Prematurity (AOP) is common, affecting the majority of infants born <34 weeks gestational age (GA). Apnea is accompanied by intermittent hypoxia (IH), which contributes to multiple pathologies, including retinopathy of prematurity (ROP), sympathetic ganglia injury, impaired pancreatic islet cell and bone development, and neurodevelopmental disabilities. Standard of care for AOP/IH includes prone positioning, positive pressure ventilation, and caffeine therapy, none of which is optimal. The objective is to support breathing in premature infants by using a simple, non-invasive vibratory device placed over limb proprioceptor fibers, an intervention using the principle that limb movements facilitate breathing.

Methods Used: Premature infants (23-34 wks GA) with clinical evidence of AOP/IH were enrolled 1 week after birth. Caffeine therapy was not a reason for exclusion. Small vibration devices were placed on one hand and one foot and activated in a 6 hour ON/OFF sequence for a total of 24 hours. Heart rate, respiratory rate, oxygen saturation (SpO2), and breathing pauses were continuously collected.

DETAILED DESCRIPTION:
Aim: To study the effect of limb proprioceptive stimulation using a vibratory device on apneic events, intermittent hypoxic episodes and bradycardias in a premature infant with apnea of prematurity.

The objective is to provide support and to assist impaired ventilation and oxygenation in apnea of prematurity (AOP). Recurrent apnea and accompanying resultant intermittent hypoxic (IH) episodes are significant concerns commonly encountered in premature infants, and optimal management is a challenge to neonatologists. AOP is defined as "a pause of breathing for more than 15-20 seconds or accompanied by oxygen desaturation (SpO2<80% for>4s) and bradycardia (heart rate<2/3 of baseline for>4s), in infants born less than 37 weeks of gestation [Moriette G et al., 2010]. When these pauses are longer (> 15s), they are frequently prolonged by obstructed inspiratory efforts, most likely secondary to loss of upper airway tonic activity [Martin RJ et al., 2012]. In extremely low birth weight (ELBW) infants, the incidence of IH progressively increases over the first 4 weeks of postnatal life, followed by a plateau and subsequent decline between 6-8 weeks.

The incidence of AOP correlates inversely with gestational age and birth weight. Nearly all infants born <29 weeks gestation or <1,000 g [Robertson CM et al., 2009], 54% at 30 to 31 weeks, 15% at 32 to 33 weeks, and 7% at 34 to 35 weeks gestation exhibit AOP [Martin RJ et al]. Both animal and human evidence show that immature or impaired respiratory control and the resultant IH exposure contribute to a variety of pathophysiologic issues via pro-inflammatory and/or pro-oxidant cascade as well as cellular mechanisms, e.g., apoptosis, leading to acute and chronic morbidities (e.g. retinopathy of prematurity, altered growth and cardiovascular regulation, disrupting zinc homeostasis which hampers insulin production and there by predisposing to diabetes in later life, cerebellar injuries and neurodevelopmental disabilities) [Martin RJ et al., 2004, Pae EK et al., 2011, 2014, ].

Current standard of care for AOP includes prone positioning, continuous positive airway pressure (CPAP) or nasal intermittent positive pressure ventilation (NIPPV) to prevent pharyngeal collapse and alveolar atelectasis, and methylxanthine therapy (caffeine, theophylline), which is the mainstay of treatment of central apnea [Reher et al., 2008; Pantalitschka T et al., 2009; Moretti C et al., 2012; Henderson-Smart DJ et al., 2010]. Apart from prone positioning, none of these interventions are optimal for early development. CPAP masks will distort the bony facial structure in early development, and methylxanthine interventions pose serious questions of neural development interactions.

Hypothesis: Applying slight vibration to the limbs will reduce the number of breathing pauses, intermittent hypoxic episodes and bradycardias in apnea of prematurity.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age > 23 weeks, < 34 weeks
2. At least 1 week old at recruitment
3. Diagnosis of apnea of prematurity (AOP)
4. Caffeine treatment will not be an exclusion

Exclusion Criteria:

1. Infants with major congenital anomalies/malformations which will influence central nervous system and long-term outcomes in these infants, such as cardiac anomalies (except for Patent Ductus Arteriosus or Ventricular Septal Defect) or major neurological malformations, like meningoencephalocele, holoprosencephaly etc.
2. Neonates who have apnea from airway issues like laryngomalacia or tracheomalacia
3. Neonates with history of hypoxic ischemic encephalopathy or Grade IV intraventricular hemorrhage

Min Age: 1 Week | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-10; Primary Completion 2015-08 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kalpashri Kesavan, MBBS, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - Ronald Reagan Medical Center - UCLA, Los Angeles, California
  - Santa Monica UCLA Mecial Center, Santa Monica, California

IPD SHARING:
Plan to Share IPD: Yes
Available online as supporting information:
  http://journals.plos.org/plosone/article?id=10.1371/journal.pone.0157349#sec019

REFERENCES:
- [Result] Kesavan K, Frank P, Cordero DM, Benharash P, Harper RM. Neuromodulation of Limb Proprioceptive Afferents Decreases Apnea of Prematurity and Accompanying Intermittent Hypoxia and Bradycardia. PLoS One. 2016 Jun 15;11(6):e0157349. doi: 10.1371/journal.pone.0157349. eCollection 2016. PMID 27304988

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of Recruitment: 10/2014-2/2016 Location: Hospital
Groups:
- All Subjects: In the same subject cardiorespiratory parameters - heart rate, respiratory rate and oxygen saturation were compared during the procedure (vibration) and without procedure (no vibration). The same subject had both control and treatment periods.
  Vibration: A device providing vibrations is placed on the subject and vibration is turned on and off in a 6 hour on/off sequence. Heart rate, respiratory pauses and oxygen saturation are compared during vibration (intervention) and without vibration (no intervention) in the same subject.
Period: Overall Study
Arm/Group | All Subjects
Started | 19
Completed | 15
Not Completed | 4

BASELINE CHARACTERISTICS:
Population: Premature neonates (23 to <34 weeks gestational age) Diagnosis of apnea of prematurity
Arm/Group | All Subjects
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 19
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: weeks] — gestational age in weeks
  weeks | 28.9 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants] — Population: In one study subject, the study interventions were discontinued due to worsening of clinical status from sepsis; 3 additional subjects were excluded from the final analysis due to data acquisition issues (missing data), leaving a final sample size of 15
  participants
    United States: number analyzed (Participants) | 15
    United States | 15
Birth Weight [Mean (Standard Deviation); unit: grams] — Birth weight in grams was obtained from medical records
  grams | 1213 (510)
Oxygen use [Count of Participants; unit: Participants] — Information regarding the fraction of inspired oxygen (FiO2) was obtained along with the mode of assisted ventilation (nasal cannula, CPAP, non-invasive ventilation etc.)
  Participants | 15
Caffeine use [Count of Participants; unit: Participants] — Information was obtained from medical charts for caffeine use
  Participants | 16

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Number of Episodes of Apnea/Breathing Pauses During Intervention and Without Intervention
Description: The total number of apneas/breathing pauses will be compared during periods of vibration (intervention) to periods of no vibrations (no intervention).
Time Frame: 12 hours of intervention/12 hours of no intervention
Population: Premature neonates (29 +/- 2.5 weeks gestational age at birth), with a diagnosis of apnea of prematurity
Measure: Mean (Standard Error); unit: breathing pauses
Groups:
- No Vibration; Vibration: In the same subject cardiorespiratory parameters - heart rate, respiratory rate and oxygen saturation were compared during the procedure (vibration) and without procedure (no vibration). The same subject had both control and treatment periods.
  Vibration: A device providing vibrations is placed on the subject and vibration is turned on and off in a 6 hour on/off sequence. Heart rate, respiratory pauses and oxygen saturation are compared during vibration (intervention) and without vibration (no intervention) in the same subject.
Arm/Group | No Vibration | Vibration
Number analyzed (Participants) | 15 | 15
breathing pauses | 284.13 (41.175) | 174.27 (22.985)

2. Secondary Outcome: Change in the Total Number of Intermittent Hypoxic Episodes to <90% Lasting >5 Seconds/Episode During the Intervention and Without Intervention
Description: The total number of intermittent hypoxic episodes to <90% (pulse oximetry) lasting >5 seconds/episode will be compared during periods of vibration (intervention) to periods of no vibrations (no intervention).
Time Frame: 12 hours of intervention/12 hours of no intervention
Population: Premature neonates (29 +/- 2.5 weeks gestational age at birth), with a diagnosis of apnea of prematurity
Measure: Mean (Standard Error); unit: IH events
Arm/Group | No Vibration | Vibration
Number analyzed (Participants) | 15 | 15
IH events | 151.67 (24.286) | 109.67 (22.661)

3. Secondary Outcome: Change in the Total Number of Bradycardia Episodes (<100 Beats Per Minute (Bpm), at Least 5 Seconds Long) During Intervention and Without the Intervention
Description: The total number of bradycardia episodes to <100 bpm lasting >5 seconds/episode will be compared during periods of vibration (intervention) to periods of no vibrations (no intervention).
Time Frame: 12 hours of intervention/12 hours of no intervention
Population: Premature neonates (29 +/- 2.5 weeks gestational age at birth), with a diagnosis of apnea of prematurity
Measure: Mean (Standard Error); unit: bradycardias
Arm/Group | No Vibration | Vibration
Number analyzed (Participants) | 15 | 15
bradycardias | 50.53 (23.2) | 14.93 (5.674)

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | All Subjects
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No